CLINICAL TRIAL: NCT04561908
Title: Transcatheter Microguidewire Drilling (TMD) for Transseptal Left Atrial Access: First-in-human Use Study
Brief Title: Transcatheter Microguidewire Drilling for Transseptal Left Atrial Access
Acronym: TMD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-5
Record Dates: First submitted 2020-09-20; First posted 2020-09-24 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Heart Diseases; Atrial Septal Dilatation
Keywords: transseptal; puncture; microguidewire
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Intervention Model Description: prospective, single-center, randomized, controlled study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional transseptal puncture (Active Comparator): Under the guidance of fluoroscopy and echocardiography, transseptal puncture was performed with Brockenbrough-needle.
  Interventions: Device: Transseptal puncture with Brockenbrough-needle
- Microguidewire-assisted transseptal puncture (Experimental): The Brockenbrough needle, with transseptal dilator and sheath, was introduced into the right atrium and engaged in the fossa ovalis, which was confirmed with angiographical and echocardiographical "tenting sign". 1) the hard-end of a 0.014-inch microguidewire drilled through atrial septum through Brockenbrough-needle; 2) then the needle was advanced into left atrium over the fixed microguidewire; 3) finally the soft-end of microguidewire was introduced into left atrium/left superior pulmonary vein through Brockenbrough-needle, which was further advanced over the fixed microguidewire.
  Interventions: Device: Microguidewire-assisted transseptal puncture

INTERVENTIONS:
Device: Transseptal puncture with Brockenbrough-needle — Conventional transseptal puncture with Brockenbrough-needle
  Arms: Conventional transseptal puncture
Device: Microguidewire-assisted transseptal puncture — Microguidewire-assisted transseptal puncture (0.014-inch microguidewire)
  Arms: Microguidewire-assisted transseptal puncture

SUMMARY:
This study aims to investigate the safety and efficacy of transcatheter microguidewire drilling (TMD) for transseptal left atrial access in patients with abnormal atrial septal morphology.

DETAILED DESCRIPTION:
Despite the widespread application and decades of experience, Brockenbrough-needle transseptal puncture still risks cardiac perforations and secondary pericardial effusion/tamponade, especially in patients with abnormal atrial septal morphology. To facilitate atrial septal crossing, different methods and devices have been developed, including radiofrequency energy, excimer laser, SafeSept wire and so on. However, these are still limited by availability and cost, and the advantages might be further offset by the potential risks. In addition, these methods are performed mainly with the linear insertion technique, which might result in less forward-force to penetrate atrial septum and displacement of needle-tip. Therefore, it is necessary to develop a safe, available and low-cost transseptal procedure for these patients.

Through a Brockenbrough needle, the hard "back-end" of the microguidewire (0.014-inch) has the potential to drill through the atrial septum with ease. Compared with a standard linear insertion technique, the penetration might be improved and less force is required with the bidirectional rotation technique, and the related risks might be reduced with the modified TSP due to the thin microguidewire. After the passage of the needle, the soft-end of microguidewire can be introduced into left pulmonary superior vein, which can become a safe rail for the introduction of puncture dilator/sheath.

In this study, we examined the effectiveness and safety of microguidewire-assisted TSP for patients with complex atrial septum.

ELIGIBILITY:
Inclusion Criteria: 1) Patients with atrial septal aneurysm (a bulging of the atrial septum of at least 10 mm beyond the plane of the atrial septum into either the right or left atrium); 2) Or patients with previous multiple transseptal punctures (≧2); 3) Or patients with thickened atrial septum (thickness ≧3 mm); 4) Or patients with enlarged right atrium (≧ 6 cm) and diminished left atrium (< 3 cm); 5) Or patients with prior mitral valve surgery; 6) Or patients with atrial baffles.

Exclusion Criteria: 1) Associated atrial septal defect or patent foramen ovale; 2) Associated interrupted inferior vena cava; 3) Presence of implanted cardiac devices; 4) Echocardiographic evidence of intracardiac thrombus, mass, tumor or vegetation; 5) Thromboembolic events within the last 6 months; 6) Patients unable to grant informed, written consent.

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-04 (Actual); Primary Completion 2022-09-04 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Procedural Success | 1 Day of procedure
  Number of participants with successful transseptal left atrial access
Related-complications | 1 Day of procedure
  Pericardial effusion

SECONDARY OUTCOMES:
Transseptal Access Procedure Time | 1 Day of procedure
  Total amount of procedure time, from the beginning of the transseptal procedure until left atrium access is obtained in each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Chaowu Yan, PhD and MD, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (2):
- China (2):
  - National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences,Fuwai Hospital, Beijing, Beijing Municipality
  - Yan Chaowu, Beijing, Select A State Or Province

IPD SHARING:
Plan to Share IPD: No